CLINICAL TRIAL: NCT03533296
Title: Individualized Positive End-expiratory Pressure Evaluation Using the Intratidal Compliance-volume Profile in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H1804-101-938
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2019-11

CONDITIONS: Lung Compliance
MeSH Terms: interventions — Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children (Experimental): Children who receive elective surgery under general anesthesia and are supported by mechanical ventilation
  Interventions: Procedure: Positive end expiratory pressure (PEEP)

INTERVENTIONS:
Procedure: Positive end expiratory pressure (PEEP) — The different levels of PEEP, 5 cmH2O, 8 cmH2O and 12 cmH2O, are applied serially. Mean respiratory compliance and intratidal compliance-volume profile are evaluated.

SUMMARY:
The investigators assess the changes in respiratory compliance according to different levels of positive end expiratory pressure (PEEP) in children under general anesthesia. In addition, the investigators evaluate the intratidal compliance-volume profile at each PEEP level and determine the optimal PEEP level during anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing surgery more than 1 hour under general anesthesia
* American Society Anesthesiologist physical status I, II

Exclusion Criteria:

* History of lung resection
* History of bronchopulmonary dysplasia or respiratory distress syndrome
* Abnormalities in chest radiography
* Laparoscopic surgery
* Abdominal surgery

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Mean respiratory compliance | During 15 minutes after applying each level of PEEP
  Mean static and dynamic compliance

SECONDARY OUTCOMES:
Compliance profile | During 15 minutes after applying each level of PEEP
  We will determine Intratidal compliance-volume profile using the changes in compliance over time
  --> I, merely increasing compliance profile; IH, increasing turning into horizontal compliance profile; D, merely decreasing compliance profile; HD, horizontal turning into decreasing compliance profile; IHD, increasing turning into horizontal and further turning into decreasing compliance profile
  If compliance profile is I, the PEEP is low. On the other hand, compliance profile is D, PEEP level is considered to be high.
Airway resistance | During 15 minutes after applying each level of PEEP
  Mean airway resistance

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, PhD, Principal Investigator — Seoul National University Hospital, Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee JH, Ji SH, Lee HC, Jang YE, Kim EH, Kim HS, Kim JT. Evaluation of the intratidal compliance profile at different PEEP levels in children with healthy lungs: a prospective, crossover study. Br J Anaesth. 2020 Nov;125(5):818-825. doi: 10.1016/j.bja.2020.06.046. Epub 2020 Jul 15. PMID 32682552